CLINICAL TRIAL: NCT01972893
Title: A Randomized, Double-blind, Placebo-controlled Phase I Clinical Study to Evaluate the Safety, Tolerability, and Pharmacokinetics of ZYD1, a Selective Glucagon-like Peptide (GLP) 1 Agonist, Following Subcutaneous Administration in Healthy Volunteers.
Brief Title: A Clinical Study to Evaluate the Safety, Tolerability, and Pharmacokinetics of ZYD1, Following Subcutaneous Administration in Healthy Volunteers
Acronym: ZYD1
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Zydus Lifesciences Limited (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: ZYD1/1001; CTRI/2011/04/001684 (Other: Clinical Trial Registration India)
Record Dates: First submitted 2012-03-05; First posted 2013-10-31 (Estimated); Last update posted 2013-10-31 (Estimated); Status verified 2013-10

CONDITIONS: Type 2 Diabetes Mellitus
Keywords: Selective GLP-1 agonist
MeSH Terms: conditions — Diabetes Mellitus, Type 2

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- ZYD1 (Experimental): Tablet ZYD1 5 to 50 mg subcutaneously Once a day (OD) or BID depending upon the pharmacokinetic profile obtained in Plan I (Single dose study)
  Interventions: Drug: ZYD1
- Placebo (Placebo Comparator): Tablet Placebo 5 to 50 mg subcutaneously OD or BID depending upon the pharmacokinetic profile obtained in Plan I (Single dose study)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: ZYD1 — Plan I - Tablet ZYD1 - 0.5, 1 , 2, 5, 10, 25 and 50 mg subcutaneously OD after overnight fasting.
  Plan II - Tablet ZYD1 - 0.5, 1 , 2, 5, 10 and 25 mg subcutaneously OD after overnight fasting.
  Plan III - Tablet ZYD1 2/5 mg subcutaneously OD after overnight fasting depending on results of Plan I.
  Other Names: Selective GLP-1 agonist
  Arms: ZYD1
Drug: Placebo — Plan I - Tablet Placebo - 0.5, 1 , 2, 5, 10, 25 and 50 mg subcutaneously OD after overnight fasting.
  Plan II - Tablet Placebo - 0.5, 1 , 2, 5, 10 and 25 mg subcutaneously OD after overnight fasting.
  Plan III - Tablet Placebo 2/5 mg subcutaneously OD after overnight fasting depending on results of Plan I.
  Arms: Placebo

SUMMARY:
ZYD1 is a novel GLP-1 receptor agonist. The ZYD1 exhibits increased stability to proteolytic cleavage, especially against dipeptidyl peptidase-4 (DPP-IV).

ZYD1 is a potent antidiabetic agent without gastrointestinal side-effects. A first in human (FIH) Phase I study intends to evaluate the safety, tolerability, pharmacokinetics and pharmacodynamics of ZYD1 in normal healthy adult volunteers.

ELIGIBILITY:
Inclusion Criteria:

1. Age: 18-45 years
2. Mentally, physically, and legally eligible to give informed consent
3. Male and female volunteers weighing between 50-75 kg and 45-75 kg respectively
4. Ability to communicate effectively with the study personnel
5. Willingness to adhere to the protocol requirements
6. For gender effect study, only females with history of sterility or at least 1 year menopause or use of long acting nonhormonal contraceptive measures (e.g., intrauterine device) will be recruited.

Exclusion Criteria:

1. Presence or history of hypersensitivity to any of the active or inactive ingredients of ZYD1 formulation
2. Presence or history of pancreatitis at any time (Serum Amylase/Serum Lipase more than upper normal limit (UNL))
3. Presence or history of severe gastrointestinal disease in the last 6 months
4. Presence or history of renal insufficiency at any time (serum creatinine above the upper limit of the reference range)
5. Active liver disease and/or liver transaminases greater than 1.5 X UNL
6. Subject with personal or family history of medullary thyroid cancer
7. Subject with personal or family history of multiple endocrine neoplasia syndrome type 2
8. Subject with serum calcitonin >50 ng/L
9. History or presence of other systemic disorders or diseases (e.g., respiratory, gastrointestinal, endocrine, immunological, dermatological, neurological, psychiatric disease or any other body system involvement)
10. Abnormal bleeding time (BT), clotting time (CT), prothrombin time (PT), and activated partial prothrombin time (APTT) tests on the day of check in
11. History or presence of any medication in the last 14 days including any medication known to interact with the Cytochrome P (CYP) 450 system
12. History or presence of significant alcoholism or drug abuse within the past 1 year
13. History or presence of significant smoking (more than 10 cigarettes per day) or consumption of tobacco products (more than 10 times per day)
14. Difficulty with donating blood
15. Systolic blood pressure more than 140 mmHg and less than 100 mmHg and diastolic blood pressure more than 90 mmHg and less than 60 mmHg
16. Pulse rate less than 60/minute and more than 100/minute
17. Any clinically significant abnormal X-ray or laboratory findings during screening
18. History or presence of any clinically significant electrocardiogram (ECG) abnormalities during screening
19. Major illness and/or major surgery in last 3 months
20. Volunteers who have participated in any drug research study other than the present trial within past 3 months
21. Volunteers who have donated one unit (350 ml) of blood in the past 3 months
22. For gender effect study, female volunteers with following criteria will not be recruited:

    * History of pregnancy or lactation in the past 3 months
    * Fertile female volunteers not protected against pregnancy by adequate long-term anti-fertility device or history of less than 1 year of menopause
    * Using hormonal contraceptives
    * Using hormone replacement therapy
    * Unable to give assurance for protection against pregnancy for 3 months after the participation in this trial
    * Positive urine pregnancy test on the day of check-in

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 56 (Actual)
Dates: Start 2011-02; Primary Completion 2012-03 (Actual); Study Completion 2012-06 (Actual)

PRIMARY OUTCOMES:
To evaluate Safety and tolerability of ZYD1 | 21 days
  The safety and tolerability shall be evaluated using physical examinations, standard laboratory tests (hematology, biochemistry and urine examination), and electrocardiogram (ECG). Spontaneously reported and solicited adverse events will also be used for safety parameters.

SECONDARY OUTCOMES:
Pharmacokinetics (PK) and Pharmacodynamic (PD) effect after single and multiple subcutaneous dose administrations in healthy adult male volunteers Gender effect study. | 1. For Plan I and III - Pre-dose (before dosing), 0.5, 1, 2, 3, 4, 6 ,8, 10, 12, 24, 48, 72 and 120 hrs post dose 2. Plan II - Day 01 - Pre-dose, 1, 2, 3, 4 and 8 hours following first dosing. Day 02 to 06 - Pre-dose of each . Day 07 - Pre-dose, 1, 2, 3,
  PK parameters evaluated for Plan I and Plan III: Cmax, Tmax, Area Under Curve (AUC)0-t, AUC 0-inf, T1/2, z, Clearance(CL), Volume of distribution (Vd) Plan II: Cmin, Tmin, Cavg, % Fluctuation, Accumulation Index, Clss, Cmax, Vd or Vss
  For urine data (Plans I, II, and III):
  Amount recovered, % recovered
  The following PD parameters (Plan I-III) will be evaluated: Plasma glucose, Serum insulin, C-Peptide, Glucagon
  Gender effects: PK and PD effect in female volunteers at preselected single dose will be compared with the results of single-dose study in male volunteers.

CONTACTS AND LOCATIONS:
Overall Officials: Rajendrakumar H Jani, PhD(Medical), Study Director — Senior Vice President - Cadila Healthcare Limited; Kevinkumar Kansagra, MD, Principal Investigator — Zydus Research Centre
Locations (1):
- Zydus Research Centre, Survey No. 396/403, Opp. Sarvotam Hotel, Nr. Nova Petrochemicals, Sarkhej-Bavla N.H. No. 8A, Village : Moraiya,, Ahmedabad, Gujarat, India